CLINICAL TRIAL: NCT02180529
Title: The Effects of Methylphenidate on the Cognitive Function of Older People With Mild Cognitive Impairment: a Randomized, Placebo Controlled, Double-blind Trial.
Brief Title: The Effects of Methylphenidate on the Cognitive Function of Older People With Mild Cognitive Impairment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting difficulties
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMC0642013
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2020-06

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: methylphenidate, elderly, mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate (Experimental): On the intervention days (days 2-4) participants will undergo cognitive assessment at 9:00 in the morning, followed by the administration (at 10:30) of different doses of Ritalin (10, 20 and 30mg) every day of intervention. Two hours after taking the drug participants will be assessed cognitively by means of Mindstreams and MoCA (Montreal Cognitive Assessment).
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Participants in the control group will receive placebo. On the intervention days (days 2-4) participants will undergo cognitive assessment at 9:00 in the morning, followed by the administration (at 10:30) of Placebo every day of intervention. Two hours after taking the placebo participants will be assessed cognitively by means of Mindstreams and MoCA (Montreal Cognitive Assessment).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — On the intervention days (days 2-4) participants will undergo cognitive assessment at 9:00 in the morning, followed by the administration (at 10:30) of different doses of Ritalin (10, 20 and 30mg) every day of intervention.
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background: The increase in life expectancy and the rise in the ratio of older to younger people in the population has resulted in an increase in the number of those suffering from a decrease in cognitive ability, such as Mild Cognitive Impairment (MCI). Methylphenidate can improve cognitive ability, mainly in memory and executive function.

Working hypothesis and aims:

This study examines the effect of Ritalin treatment in older people suffering from MCI. Our hypothesis is that treatment with Ritalin will improve cognitive function in those suffering from MCI, especially in the domains of attention and executive function.

Methods A randomized, double-blind, case-control study. 120 patients older than 65 years of age diagnosed as suffering from MCI in the past year in geriatric assessment facilities in Beersheva. Patients will be randomized in equal groups to either the study group (Ritalin treatment) and control group (placebo). Each participant will attend the geriatric unit for four consecutive days: on the day prior to beginning the intervention participants will undergo cognitive assessment at 9:00 am. On the intervention days (days 2-4) participants will undergo cognitive assessment at 9:00 in the morning, followed by the administration (at 10:30) of different doses of Ritalin (10, 20 and 30mg) every day of intervention. Participants in the control group will receive placebo. Two hours after taking the drug or placebo participants in both groups will be assessed cognitively by means of Mindstreams and MoCA (Montreal Cognitive Assessment).

Expected results: Ritalin treatment will improve the cognitive function of the subjects, mainly in the domains of concentration and executive function

ELIGIBILITY:
Inclusion Criteria:

* >65 years old
* Male and Female
* Living in the community

Exclusion Criteria:

* Suffer from unstable conditions, for example, unstable heart disease, severe heart failure, severe renal failure, cirrhosis, blood pressure above 160/100;
* patient who suffer from glaucoma, hyperthyroididsm, epilepsy, patients after stroke, patient with Parkinson's disease, major depression, schizophrenia or receiving neuroleptic drugs;
* patient who suffer from dementia
* patients that recieve treatment in acetylcholinesterase inhibitors or memantine.
* known sensitivity to methylphenidate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
cognitive function | Twice a day during 3 days
  Each participant will attend the geriatric unit for four consecutive days: on the day prior to beginning the intervention participants will undergo cognitive assessment at 9:00 am. On the intervention days (days 2-4) participants will undergo cognitive assessment at 9:00 in the morning, followed by the administration (at 10:30) of different doses of Ritalin (10, 20 and 30mg) every day of intervention. Participants in the control group will receive placebo. Two hours after taking the drug or placebo participants in both groups will be assessed cognitively by means of Mindstreams and MoCA (Montreal Cognitive Assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Press, M.D, Principal Investigator — dr.
Locations (1):
- Clalit Health Service, Beersheba, Israel